CLINICAL TRIAL: NCT00356928
Title: Cyclophosphamide Plus Transplantation of Partially HLA-mismatched (Haploidentical), CD8+ T Cell-depleted Peripheral Blood Cells for Patients With Myelodysplastic Syndrome, Acute Myeloid Leukemia, Lymphoma, or Myeloproliferative Disorders
Brief Title: Cyclophosphamide Plus T-Cell Transplantation for Patients With Hematologic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0551; R21CA121588 (NIH); P30CA006973 (NIH); NA_00000901 (Other: JHMIRB)
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; secondary acute myeloid leukemia; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cyclophosphamide + T cells (Experimental): Conditioning regimen with cyclophosphamide followed by donor T cells on Day 0.
  Interventions: Drug: Cyclophosphamide; Biological: Donor T cells

INTERVENTIONS:
Drug: Cyclophosphamide — 50 mg/kg/day intravenously (IV) on Days -2 and -1.
  Other Names: Cytoxan; Cy; CTX
Biological: Donor T cells — CD8-depleted T cells given IV on Day 0. Dose levels are as follows (all doses in cells/kg):
  Dose level 1: 1E5 CD4+ cells and less than 3.2E3 CD8+ cells Dose level 2: 1E6 CD4+ cells and less than 3.2E4 CD8+ cells Dose level 3: 1E7 CD4+ cells and less than 3.2E5 CD8+ cells Dose level 4: 5E7 CD4+ cells and less than 1.6E6 CD8+ cells

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of abnormal blood cells, either by killing the cells or by stopping them from dividing. Giving cyclophosphamide together with donor lymphocytes that have been treated in the laboratory may be an effective treatment for myelodysplastic syndromes or myeloproliferative disorders.

PURPOSE: This clinical trial is studying the best dose of donor lymphocytes when given together with cyclophosphamide in treating patients with myelodysplastic syndromes or myeloproliferative disorders.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of allogeneic CD8-positive T-cell-depleted, haploidentical donor lymphocytes when given after cyclophosphamide in patients with myelodysplastic syndromes or myeloproliferative disorders.

OUTLINE: Patients receive cyclophosphamide on days 1 and 2. Patients then undergo infusion of allogeneic T-cell depleted donor lymphocytes on day 3.

Cohorts of patients receive escalating doses of CD8-positive T-cell-depleted haploidentical donor lymphocytes until the maximum tolerated dose is determined.

PROJECTED ACCRUAL: A total of 44 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Myelodysplastic syndromes (MDS)

    * International Prognostic Scoring System (IPSS) score ≥ intermediate-2
  * Chronic myelomonocytic leukemia
  * Acute myeloid leukemia arising from MDS
* Must have failed or are ineligible for or intolerant to treatment with azacitidine

  * Patients with normal marrow cytogenetics or an isolated 5q- abnormality must have failed or are ineligible for or intolerant to treatment with lenalidomide
  * Patients who are HLA-DR15-positive must have failed or are ineligible for pharmacologic immunosuppression (e.g., anti-thymocyte globulin, cyclosporine, steroids)
* No presence of cytotoxic antibodies against donor lymphocytes
* No HLA-identical donor available OR ineligible for HLA-identical allogeneic bone marrow transplantation
* HLA partially mismatched (haploidentical) related donor available

  * First-degree related donor, including half-siblings or first cousins
  * Inherited recombinant haplotype from parents allowed if donor shares ≥ 1 HLA antigen at each of the HLA-A, -B, and DR loci

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 OR Karnofsky PS 80-100%
* Bilirubin < 3.0 mg/dL
* AST and ALT ≤ 4 times upper limit of normal
* Creatinine < 3.0 mg/dL
* LVEF > 35%

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* No prior transfusions from donor
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) or radiotherapy
* No other concurrent investigational drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of haploidentical donor lymphocytes | 60 days
  Maximum dose in cells per kilogram that did not cause dose-limiting toxicity (defined as grade 3-5 non-hematologic toxicity, death within 60 days related to protocol treatment, aplasia related to treatment, or grade 3-4 graft-vs-host-disease).

SECONDARY OUTCOMES:
Disease response | Up to 6 months
  Percentage of participants who had a complete remission after protocol treatment.
Duration of response | Up to 6 months
  Median length of response (in months) of participants who had a complete remission after protocol treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yvette L. Kasamon, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No